CLINICAL TRIAL: NCT01387126
Title: A Randomized, Controlled Trial Evaluating the Effects of a High Viscosity Dietary Fibre, as Part of a Medically Supervised Weight Management Program, on Body Weight in Overweight and Obese Individuals
Brief Title: Effects of a High Viscosity Dietary Fibre, as Part of a Medically Supervised Weight Management Program
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No grant funding for this trial.
Sponsor: Canadian Center for Functional Medicine (Other)
Collaborators: University of British Columbia (Other); InovoBiologic Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 004
Record Dates: First submitted 2011-06-30; First posted 2011-07-04 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2017-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

ARMS (2):
- Novel fibre supplement (Experimental): The full dose of the study intervention is 15 grams per day.
  Interventions: Dietary Supplement: Novel fibre supplement
- Weight management program (No Intervention)

INTERVENTIONS:
Dietary Supplement: Novel fibre supplement — The full dose of the study intervention is 15 grams per day.
  Arms: Novel fibre supplement

SUMMARY:
The aim of this study is to investigate whether the supplementation of a medically supervised weight management program with a novel fibre supplement, improves body weight, body composition, and laboratory measurements in overweight and obese individuals. All subjects will participate in the medical weight management program however the intervention group will have 5 grams of a novel fibre supplemented to each meal while the control group will not.

ELIGIBILITY:
Inclusion Criteria:

* BMI 27 - 30 Kg/m2 with 1 weight-related comorbidity and/or BMI 30 - 50 Kg/m2
* Ability to provide written informed consent in accordance with Good Clinical Practice (GCP) and local legislation in English

Exclusion Criteria:

* Medications and supplements that affect body weight and appetite
* Type 2 diabetes on insulin treatment
* Contraindications to low calorie diet
* Any allergies to study product ingredients
* Any other medical, social or geographic condition, which, in the opinion of the investigator would not allow safe completion of the protocol.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Body weight | 52 weeks

SECONDARY OUTCOMES:
Body composition | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Lyon, MD, Principal Investigator — Canadian Centre for Functional Medicine
Locations (1):
- Canadian Centre for Functional Medicine, Coquitlam, British Columbia, Canada